CLINICAL TRIAL: NCT04033315
Title: User Performance of the L-PLUS Blood Glucose Monitoring System
Brief Title: Performance of the L-PLUS BGMS by Persons With Diabetes Mellitus
Status: Completed | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-PRO-2019-002-01
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; BGMS; blood glucose monitoring system; fingerstick; AST self-test; YSI Glucose Analyzer
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: All subjects will be assigned to use the L-PLUS meter
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Untrained Subjects with Diabetes use the L-PLUS BGMS (Experimental): Untrained subjects with Diabetes test capillary fingerstick and palm blood (and study staff test subject fingerstick blood) using the L-PLUS BGMS. All blood glucose results are compared to reference method results obtained with subject capillary plasma. Also, study staff test venous blood and blood glucose results are compared to reference method results obtained from subject venous plasma.
  Interventions: Device: L-PLUS meter

INTERVENTIONS:
Device: L-PLUS meter — Blood Glucose Monitoring System

SUMMARY:
L-PLUS (Lightning PLUS) is the code name of a blood glucose monitoring system (BGMS) consisting of a new meter and marketed CONTOUR PLUS® test strip. This clinical trial will assess the performance (accuracy) of the L-PLUS meter by lay users with diabetes enrolled as subjects in the study, and by health care professionals (also called study staff).

The trial will follow the requirements and procedures described in ISO 15197:2013 International Standard.

DETAILED DESCRIPTION:
This study is designed to satisfy the ISO 15197:2013, Section 8 requirements.

The study will be conducted at a minimum of one clinical site and enroll a total of approximately 130 persons with diabetes.

For this study, there must be at least 120 evaluable results each for fingerstick and AST self-test results, as well as for staff testing subject fingertip and venous blood using the L-PLUS BGMS. Subject enrollment will continue until the required evaluable samples are collected.

The subjects will be 18 years and older. Each subject will make one visit, lasting approximately 1 hour at the clinical site. All subjects will complete the informed consent process before performing any study procedures.

All Subjects will be assigned a L-PLUS meter and one Contour Plus test strip lots. The untrained subjects will learn to use the L-PLUS meter by reading the instructional materials. Each subject will perform one fingerstick self-test, one palm test, and staff will perform a fingerstick test on the subject.

Subjects will be given a venipuncture and the venous blood will be tested by the study staff with the L-PLUS system. All subject capillary and AST self-test results and study staff fingerstick results will be compared to YSI fingerstick results. Venous blood meter tests will be compared to YSI results of the corresponding venous blood. Hematocrit will be measured for all subjects. All Subjects will then complete a questionnaire (Questionnaire 1) to provide feedback on the meter system and instructions for use.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* People with diabetes (PWD) - type 1 or type 2
* Ability to speak, read and understand English. Subjects must demonstrate ability to read a paragraph from the first page of the UG to qualify for the study.
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy (self-reported)
* Physical, visual or neurological impairments that would make the person unable to perform testing with the BGMS.
* Previous participation in a blood glucose monitoring study using the Ascensia's Contour Next (Lightning Next) and Lightning PLUS (L-PLUS or Contour Plus ELITE) BGMS.
* Working for a medical laboratory, hospital or other clinical setting that involves training on or clinical use of blood glucose monitors.
* Being in this trial during or less than two days since xylose absorption testing (Xylose in the blood is known to cause interference).
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company.
* A condition, which in the opinion of the investigator or designee, would put the person or study conduct at risk. The reason for exclusion will be clearly documented by investigator or designee on the subject disposition form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rainier Clinical Research Center, Inc., Renton, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Untrained Subjects With Diabetes Use the L-PLUS BGMS
Started | 130
Completed | 129
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Untrained Subjects With Diabetes Use the L-PLUS BGMS
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 106
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 115
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 31
  White | 72
  More than one race | 3
  Unknown or Not Reported | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of BGMS Compared to the Reference Analyzer - Fingerstick Blood Test
Description: Accuracy of BGMS test with fingerstick blood. The results of the fingerstick meter test performed by the participant will be compared to results of the same blood on a laboratory reference analyzer using pre-specified accuracy criteria.
Time Frame: Day 1
Population: Persons with diabetes perform finger stick tests.
Measure: Count of Participants; unit: Participants
Arm/Group | Untrained Subjects With Diabetes Use the L-PLUS BGMS
Number analyzed (Participants) | 128
Participants | 127

2. Secondary Outcome: Accuracy of BGMS Compared to the Reference Analyzer - Palm Alternative Site Test (AST)
Description: Accuracy of BGMS test with palm blood. The results of the palm blood meter test performed by the participant will be compared to results of the same blood on a laboratory reference analyzer using pre-specified accuracy criteria
Time Frame: Day 1
Population: Persons test their blood from palm.
Measure: Count of Participants; unit: Participants
Arm/Group | Untrained Subjects With Diabetes Use the L-PLUS BGMS
Number analyzed (Participants) | 121
Participants | 119

3. Secondary Outcome: Accuracy of BGMS Compared to the Reference Analyzer - Venous Blood
Description: Accuracy of BGMS using venous blood compared to the reference analyzer for all subjects using pre-specified accuracy criteria
Time Frame: Day 1
Population: Venous blood is tested on each participant.
Measure: Count of Participants; unit: Participants
Arm/Group | Untrained Subjects With Diabetes Use the L-PLUS BGMS
Number analyzed (Participants) | 129
Participants | 129

ADVERSE EVENTS:
Time Frame: Day 1
Arm/Group | Untrained Subjects With Diabetes Use the L-PLUS BGMS
All-Cause Mortality (participants affected / at risk) | 0/130
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 0/130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT04033315/Prot_SAP_000.pdf